CLINICAL TRIAL: NCT03086564
Title: A Basic-clinical Translational Research in Hepatitis B Virus (HBV)-Specific Antigen Peptides and HepG2 Cell Lysate Co-activated Dendritic Cells Combined With Transarterial Chemoembolization (TACE) in HBV-related HCC Treatment
Brief Title: A Basic-clinical Translational Research in Hepatitis B Virus (HBV)-Specific Antigen Peptides and HepG2 Cell Lysate Co-activated Dendritic Cells Combined With Transarterial Chemoembolization (TACE) in HBV-related HCC Treatment (BTRHBVAPHCLCDCCTCHBVHCCT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuehua Huang (Other)
Responsible Party: Sponsor-Investigator, Yuehua Huang, Director, Provincial Key Laboratory of Liver, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: huangyuehuateam
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; ADCC; TACE; immuno therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Antibody-Dependent Cell Cytotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADCC & TACE (Experimental): The first course :
  Patients in the first day of a clinical course will be performed TACE solely and keep 40ml blood sample as baseline sample for scientific research;in the 17th day, 10ml blood will be taken to culture activated dendritic cells;in 29th day, cyclophosphamide(CY) 250mg/m2 is used through an intravenous drip;in 31th day,patients are going to be performed TACE,1-2*10^8 activated dendritic cells are dripped through peripheral vein, 40ml blood sample will be taken for clinical research, simultaneously.
  The 31th day in the first course is the same as the first day of the second course, then we come to next therapy course.
  31 days are a course of treatment, health conditions of patients who participate in will be monitored closely in the process. After previous 3-courses followed-up period, one course will be changed into 93 days.
  Interventions: Biological: ADCC & TACE
- TACE (Active Comparator): Every course:
  In the first day,patients are performed TACE solely and taken 40ml blood as baseline sample for scientific research;in the 29th day,patients are needed to reach hospital to check related indicators. In the 31th day, patients are performed TACE again.
  The 31th day is the same as the first day in the second course.
  31 days are a course of treatment, health conditions of patients who participate in will be monitored closely in the process. After previous 3-courses followed-up period, one course will be changed into 93 days.
  Interventions: Procedure: TACE

INTERVENTIONS:
Biological: ADCC & TACE — Experimental groups will be given TACE as well as Activated-Dendritic Cells(1-2*10^8,intravenous drip),simultaneously.Cyclophosphamide(250mg/cm2,intravenous drip) will be used two days before TACE performed.
  Arms: ADCC & TACE
Procedure: TACE — TACE solely in the first day of a clinical course.
  Arms: TACE

SUMMARY:
The effect of anti-tumor treatment is not satisfying in HBV-related hepatocellular carcinoma (HBV-HCC) for reasons that HBV-HCC carries highly heterogeneous antigens to facilitate cancer cells escaping from immune surveillance and constructs an immunosuppressive microenvironment. Correspondingly, dendritic cells activated by HBV antigen peptides and HepG2 cell protein lysate can efficiently present T cells with antigens of HCC to sensitize their antitumor properties meanwhile cyclophosphamide(CY) can effectively improve the microenvironment of immunity. Therefore, we put forward a new scientific therapy called "Activated Dendritic-cells Combined Cyclophosphamide" (ADCC) combining with TACE for patients with advanced hepatocellular carcinoma to prolong their survival time.

DETAILED DESCRIPTION:
Patients who have good compliance complying with the inclusion criteria will be enrolled into our research. The 70 patients will be randomly assigned to experimental group and control group with the ratio of 1:1, one group (control group) will go on receiving the TACE treatment solely; another group (experimental group) after enrollment will receive TACE in the first course.Then 10ml blood is taken for activated dendritic cells culture.CY treatment will be performed on patients in reasonable dose two days before the second TACE.The day when the second TACE performed, these patients will receive activated-dendritic cells simultaneously. 31 days after the first TACE therapy, all patients are determined if they should continue an additional course by monitoring their blood parameters, tumor indicators and imaging examinations. Additionally, we are setting up a treatment course containing 31 days and going to change one course into 93 days after the third course.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients with history of hepatitis B infection
  * Stage B or C in Barcelona Clinic Liver Cancer(BCLC)
  * Eastern Cooperative Oncology Group(ECOG) scores <= 2.(without portal vein involved)
  * Patients have been unable to be performed surgery or liver transplant
  * Patients are appropriate to be performed TACE
  * 18 or over 18 years old
  * Patients haven't received radiation therapy or chemotherapy or immunotherapy
  * Normal renal function
  * Blood routine test:Hb>=9g/L,white cell count>=1.5*10^9/L,platelet count>=50*10^9
  * Liver function: bilirubin<=50ummol/L,aspartate aminotransferase (AST) or alanine aminotransferase (ALT)<=5 times the upper limit of normal
  * Child-Pugh score<=9
  * Human Chorionic Gonadotropin (HCG) test negative(-) if patients are women of reproductive ages
  * Women of reproductive ages promise to contracept until therapy course has been finished for 3 months
  * Patients who have signed up informed consents
* Exclusion Criteria:

  * Extrahepatic metastasis of hepatocellular carcinoma
  * History of embolism, chemotherapy or radiation
  * History of major surgery in last 4 weeks
  * History of radiofrequency ablation in last 6 weeks
  * Acute infections in last 2 weeks
  * Child-Pugh scores>9
  * Patients with hepatic encephalopathy
  * Patients with ascites needed drainage
  * HCC with portal vein involved
  * Patients have history of cancer
  * Patients have history of HIV
  * Pregnant women
  * Patients with severe diseases like cardiac dysfunction
  * Patients with mental illness that influence signing informed consents
  * HBV infection combined with other types of hepatitis
  * Patients with autoimmune diseases
  * Immunosuppressant drugs users
  * Patients cannot follow our trial principle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Imaging signs | 4 years
  The size of tumor decrease.
Alpha-fetoprotein (AFP) | 4 years
  To decrease AFP to a low level
Glypican-3 | 4 years
  To decrease Glypican-3 to a low level

CONTACTS AND LOCATIONS:
Overall Officials: Lubiao Chen, Dr., Study Chair — the third affiliated hospital of sun yet-sen university
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China